CLINICAL TRIAL: NCT04599660
Title: Follow-up in Low Risk Gastrointestinal Stromal Tumors (GISTs) - Retrospective Analysis of Clinical Features and Outcomes
Brief Title: Study in Low Risk Gastrointestinal Stromal Tumor (GISTs)
Acronym: RetroGIST
Status: Completed | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG-RetroGIST LR
Record Dates: First submitted 2020-10-15; First posted 2020-10-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-12

CONDITIONS: GIST
Keywords: GIST; Gastro Intestinal Stromal Tumor
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Risk GISTs: This cohort include patients affected by primary GIST at very-low and low risk of recurrence/progression, referred to participating Institutions between January 2000 and February 2020.
  Interventions: Other: Treatment of Low Risk GISTs according clinical practice (includes drugs, surgery or any other received treatments)

INTERVENTIONS:
Other: Treatment of Low Risk GISTs according clinical practice (includes drugs, surgery or any other received treatments) — This observational study collects all the treatments received by the patients according clinical practices or experimental trials and therefore includes drug/biological/surgical and any other applicable treatments

SUMMARY:
This is a multi-institutional retrospective study in order to identify the most relevant and advisable features of follow-up, and to explore its impact on principal clinical outcomes. Moreover, a dedicated effort will be pursued to identify the peculiar characteristics (if any) of patients that experienced recurrence of the disease.

The study will collect data about patients affected by primary GIST at very-low and low risk of recurrence/progression, referred to participating Institutions between January 2000 and February 2020

DETAILED DESCRIPTION:
In the field of soft tissue sarcomas, Gastrointestinal Stromal Tumors (GIST) represents a really peculiar neoplasm for its biological and clinical properties. Surgery (if feasible) is the main therapeutic approach for all the patients with localized disease, while a pharmacological adjuvant treatment is reserved to those with a relevant risk of recurrence/progression.

After tumor removal, clinical and radiological follow-up is of central importance to early intercept recurrence and to evaluate the most correct subsequent therapeutic approach. In particular, for the group of patients with GIST at very-low and low risk of recurrence/progression, the evidences to support a specific follow-up program and its features are poor.

On the basis of the aforementioned considerations, we propose a multi-institutional retrospective study in order to identify the most relevant and advisable features of follow-up, and to explore its impact on principal clinical outcomes. Moreover, a dedicated effort will be pursued to identify the peculiar characteristics (if any) of patients that experienced recurrence of the disease.

The study will collect data about patients affected by primary GIST at very-low and low risk of recurrence/progression, referred to participating Institutions between January 2000 and February 2020

ELIGIBILITY:
Inclusion Criteria:

* >18 years at diagnosis
* primary GIST removed by surgery or endoscopic procedures
* availability of medical data needed for the study
* very-low and low risk GIST defined as:

  * largest size of < 3 cm (for all sites of origin)
  * gastric GIST with ≤ 5/50 High Power Fields (HPF) mitoses and ≤ 10 cm in the largest size
  * gastric GIST with > 5/50 HPF mitoses and ≤ 5 cm in the largest size
  * intestinal GIST with ≤ 5/50 HPF mitoses and ≤ 5 cm in the largest size

Exclusion Criteria:

* Metastases at diagnosis.
* Previous treatment with imatinib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by primary GIST at very-low and low risk of recurrence/progression, referred to participating Institutions between January 2000 and February 2020.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
To describe the most relevant features of follow-up in very-low and low risk GIST patients | Change from diagnosis (baseline)
  Collection of retrospectively imaging characteristics
To describe the most relevant features of follow-up in very-low and low risk GIST patients | At 1 year
  Collection of retrospectively imaging characteristics.
To describe the most relevant features of follow-up in very-low and low risk GIST patients | At 2 years
  Collection of retrospectively imaging characteristics.
To describe the most relevant features of follow-up in very-low and low risk GIST patients | At 3 years
  Collection of retrospectively imaging characteristics.
To describe the most relevant features of follow-up in very-low and low risk GIST patients | At 5 years
  Collection of retrospectively imaging characteristics.
To evaluate the onset of other neoplasms in very-low and low risk GIST patients | Chage from baseline (time of diagnosis) at 5 years
  Onset of other neoplasm will be recoreded

SECONDARY OUTCOMES:
To assess baseline clinical and disease-specific factors with possible impact on survival analyses. | Every 3 months (Month 3, Month 6, Month 9...) up to 5 years
  Collection of clinical symptoms, pathological and molecular characteristics at disease presentation/diagnosis
Recurrence-free survival (RFS) | Every 3 months (Month 3, Month 6, Month 9...) up to 5 years
  Time elapsed form the treatment (any) start and the onset of recurrence
Post-recurrence progression-free survival (PR-PFS) | Every 3 months (Month 3, Month 6, Month 9...) up to 5 years
  Time elapsed form the onset of 1st progression to a further progression
Disease-Specific survival (DSS) | at 5 years
  Time elapsed for the diagnosis to the death of disease
Overall survival (OS). | at 5 years
  Time elapsed for the diagnosis to the death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Grignani, Study Chair — giovanni.grignani@ircc.it
Locations (13):
- Italy (13):
  - Azienda Ospedaliero-Universitaria Di Bologna, Bologna, BO
  - Nuovo Ospedale di Prato, Prato, Firenze
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Ospedale San Giovanni Bosco, Torino, TO
  - Policlinico S.Orsola Malpighi - Unit of Medical Oncology, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS INT Milano, Milan
  - Istituto Nazionale Tumori Regina Elena - Unit of Medical Oncology I, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joensuu H, Hohenberger P, Corless CL. Gastrointestinal stromal tumour. Lancet. 2013 Sep 14;382(9896):973-83. doi: 10.1016/S0140-6736(13)60106-3. Epub 2013 Apr 24. PMID 23623056
- [Background] Gold JS, Gonen M, Gutierrez A, Broto JM, Garcia-del-Muro X, Smyrk TC, Maki RG, Singer S, Brennan MF, Antonescu CR, Donohue JH, DeMatteo RP. Development and validation of a prognostic nomogram for recurrence-free survival after complete surgical resection of localised primary gastrointestinal stromal tumour: a retrospective analysis. Lancet Oncol. 2009 Nov;10(11):1045-52. doi: 10.1016/S1470-2045(09)70242-6. Epub 2009 Sep 28. PMID 19793678
- [Background] D'Ambrosio L, Palesandro E, Boccone P, Tolomeo F, Miano S, Galizia D, Manca A, Chiara G, Bertotto I, Russo F, Campanella D, Venesio T, Sangiolo D, Pignochino Y, Siatis D, De Simone M, Ferrero A, Pisacane A, Dei Tos AP, Aliberti S, Aglietta M, Grignani G. Impact of a risk-based follow-up in patients affected by gastrointestinal stromal tumour. Eur J Cancer. 2017 Jun;78:122-132. doi: 10.1016/j.ejca.2017.03.025. Epub 2017 Apr 24. PMID 28448856
- [Background] Joensuu H, Reichardt P, Eriksson M, Sundby Hall K, Vehtari A. Gastrointestinal stromal tumor: a method for optimizing the timing of CT scans in the follow-up of cancer patients. Radiology. 2014 Apr;271(1):96-103. doi: 10.1148/radiol.13131040. Epub 2013 Nov 18. PMID 24475826
- [Background] Rossi S, Miceli R, Messerini L, Bearzi I, Mazzoleni G, Capella C, Arrigoni G, Sonzogni A, Sidoni A, Toffolatti L, Laurino L, Mariani L, Vinaccia V, Gnocchi C, Gronchi A, Casali PG, Dei Tos AP. Natural history of imatinib-naive GISTs: a retrospective analysis of 929 cases with long-term follow-up and development of a survival nomogram based on mitotic index and size as continuous variables. Am J Surg Pathol. 2011 Nov;35(11):1646-56. doi: 10.1097/PAS.0b013e31822d63a7. PMID 21997685
- [Background] Casali PG, Abecassis N, Aro HT, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Brodowicz T, Broto JM, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kasper B, Kopeckova K, Krakorova DA, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee and EURACAN. Gastrointestinal stromal tumours: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv267. doi: 10.1093/annonc/mdy320. No abstract available. PMID 30188977